CLINICAL TRIAL: NCT01321580
Title: Comparison of the Hemoglobin Results Obtained With the Masimo Pronto 7 and the Clinical Laboratory Measurement Study
Brief Title: Hemoglobin MASIMO (Pronto 7) and Laboratory Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/43; 2010-A00541-38 (Other: ANSM)
Record Dates: First submitted 2011-03-19; First posted 2011-03-23 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group A (Experimental)
  Interventions: Device: Masimo Pronto 7

INTERVENTIONS:
Device: Masimo Pronto 7 — non invasive hemoglobin determination by the Masimo Pronto 7 versus laboratory hemoglobin measurement

SUMMARY:
The purpose of this study is to compare the hemoglobin results obtained with the Masimo Pronto 7 and the Clinical Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* emergency unit patients requiring an hemoglobin determination

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
accuracy of Masimo Pronto 7 | 6 months
  correlation, Bland and Altman analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Foch, Suresnes, France

REFERENCES:
- [Derived] Gayat E, Aulagnier J, Matthieu E, Boisson M, Fischler M. Non-invasive measurement of hemoglobin: assessment of two different point-of-care technologies. PLoS One. 2012;7(1):e30065. doi: 10.1371/journal.pone.0030065. Epub 2012 Jan 6. PMID 22238693